CLINICAL TRIAL: NCT00818467
Title: 3% Dihydroxyacetone (DHA or Sunless Tanning Agent) Inhibits Vitamin D Production in the Skin in Response to Ultraviolet Light
Brief Title: UVB Light and Sunscreen
Acronym: Sunscreen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: The UV Foundation (Other)
Responsible Party: Laura Armas, Creighton University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Creighton 7
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Vitamin D Status
Keywords: Skin tone; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tanning spray (Experimental): To characterize the 25(OH)D response to 4 weeks of thrice weekly 40 mJ of UV-B light in a group of normal subjects with skin types I and II while using multiple applications of 3% DHA for five weeks.
  Interventions: Other: Tanning spray
- UVB (Active Comparator): To characterize the 25(OH)D response to 4 weeks of thrice weekly 40 mJ of UV-B light in a control group of normal subjects with skin types I and II who are not using 3% DHA applications.
  Interventions: Other: UVB

INTERVENTIONS:
Other: Tanning spray — using 3% DHA twice a week for the 1st week and then once a week for 4 weeks and receiving 40mJ UV-B phototherapy three times a week for four weeks
  Arms: Tanning spray
Other: UVB — receiving 40mJ UV-B phototherapy three times a week for four weeks
  Arms: UVB

SUMMARY:
Patients need vitamin D which is normally produced in the skin in response to ultraviolet light from the sun. Vitamin D is important for calcium absorption and good bone health. Physicians have been using sunscreens to protect patients from skin cancer and the aging effects of sunlight for a least a half a century. Dermatologists have promoted sunscreen use to restrict sunlight exposure especially in white Caucasians. If this behavior is done 100% of the time when outdoors individuals may suffer from vitamin D deficiency. It is impossible to influence persons' behavior to wear sunscreens all the time when outdoors. With the use of sunless tanning agent (DHA), once a week, we can obtain a continuous sunscreen in the top layer of the skin that will not wash off, can't be removed with soap and water, or removed by perspiration. Under these circumstances we can answer the scientific question, will sunscreen use inhibit the production of vitamin D in the skin?

ELIGIBILITY:
Inclusion Criteria:

* males or females
* ages 19-50 with less than 16 oz milk per day
* less than 10 hours of sun per week
* no Vitamin D supplements
* no anticonvulsants
* no barbiturates
* no steroids
* no meds that increase photosensitivity
* no granulomatous disease
* no liver or kidney disease
* no history of skin cancer
* BMI less than 30
* skin types I & II

Exclusion Criteria:

* None

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2008-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To measure the response of 25(OH)D to 40 milliJoules of UV-B light in white Caucasians with melanoidins-sunscreen from 3% DHA in comparison to the response of control subjects who have not used 3% DHA. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Armas, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States